CLINICAL TRIAL: NCT00283634
Title: A Randomized, Non-comparative, Multicenter, Open-Label, Phase 2 Study of Tarceva™ (Erlotinib) Alone and of Tarceva Plus VELCADE* (Bortezomib) for Injection in Patients With Relapsed or Refractory, Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Tarceva for Use in Patients With Relapsed or Refractory Metastatic Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient efficacy
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C05005
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: NSCLC
MeSH Terms: interventions — Erlotinib Hydrochloride; Bortezomib

INTERVENTIONS:
Drug: erlotinib and bortezomib

SUMMARY:
Tarceva, an orally available small molecule, has demonstrated potent activity in tumor models and humans. This randomized, open-label phase 2 study of Tarceva alone and of Tarceva plus VELCADE is designed primarily to determine the objective tumor response rates to these treatments in patients with Stage IIIB or Stage IV non-small cell lung cancer (NSCLC) that is refractory to or has relapsed after front-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1)Relapsed or refractory, Stage IIIB or Stage IV NSCLC that has been histologially or cytologically confirmed. 2)One prior line of conventional cytotoxic chemotherapy. 3)Documented progressive disease(PD) during or since last prior therapy as determined by the investigator. 4)18 y/o or older. 5)Have measurable disease by RECIST. 6)Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1. 7)Life expectancy greater than 3 mo from the date of enrollment. 8)Female patient is either post-menopausal, surgically sterilized or willing to use an acceptable method of birth control. 9)Male pateint agrees to use an acceptable method of birth control during study treatment. 10)Provide written informed consent before the conduct of any study-related procedure. 11)Willing and able to comply with the protocol requirements.

Exclusion Criteria:

1)Previous treatment w/VELCADE. 2)Pre-existing interstitial lung disease. 3)Peripheral neuropathy of Grade 2 or greater. 4)Diarrhea or vomiting greater than Grade 1 in intensity whether in the absence or presence of antidiarrheal and/or antiemetic therapy. 5)Chemotherapy, radiation therapy, treatment wtih monoclonal Antibodies, or major surgery w/in 4 wks prior to enrollment. 6)Documented greater than 10% WT loss in the 6 wks. prior to enrollment. 7)Inadequate organ function during screening as per laboratory values. 8)Myocardial infarction w/in 6 months prior to enrollment. 9)Brain metastases. 10)Any malignancy other than NSCLC occuring w/in 5 years of enrollment with the exception of basal cell carcinoma of the sin, and carcinoma in situ of the cervix. 11)Hx of allergic reaction to compounds containing boron or mannitol. 12)Known human immunodeficiency virus (HIV)+ or hepatitis B. 13)Poorly controlled hypertension, diabetes mellitus, or pyschiatric illness. 14)Pregnant or breast-feeding woman. Confirmation that patient is not pregnant must be established by a negative serum (B-hCG).15)Currently enrolled in another clinical research study or has received an investigational agent w/in 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-08; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennesee, Knoxville, Tennessee, United States